CLINICAL TRIAL: NCT06005311
Title: A Randomized Double-blind Controlled Study of the Cumulative Live Birth Rate of IVF Following Sperm Preparation by Microfluidic Chip Method Versus Density-gradient Centrifugation Method
Brief Title: Microfluidic Chip Method Versus Density-gradient Centrifugation Method in IVF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Ernest Hung-Yu Ng (Other)
Responsible Party: Sponsor-Investigator, Professor Ernest Hung-Yu Ng, Clinical Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW 23-293
Record Dates: First submitted 2023-06-29; First posted 2023-08-22 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Infertility
Keywords: microfluidic chip; density-gradient centrifugation; in-vitro fertilisation; sperm preparation
MeSH Terms: conditions — Infertility | interventions — Centrifugation, Density Gradient

STUDY DESIGN:
Intervention Model Description: Infertile patients attending IVF treatment at the Centre of Assisted Reproduction and Embryology, Queen Mary Hospital and Kwong Wah Hospital will be recruited during ovarian stimulation for IVF. Subsequently, they will be randomly assigned on the day of oocyte retrieval by a laboratory staff into one of the following two groups: (1) the microfluidic chip group and (2) the density gradient group for sperm preparation and subsequent use in fertilization. Other IVF procedures will be the same as our usual practice.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both patients and clinicians were blinded from the group allocation i.e. a double blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- microfluidic chip method (Experimental): Microfluidic chip method has been used for sperm sorting in order to select the most motile and morphologically normal sperm for use in assisted reproductive technologies (ART) such as in vitro fertilization (IVF) and intracytoplasmic sperm injection (ICSI).
  In the microfluidic chip method for sperm sorting, a small amount of semen sample is loaded onto the chip, which contains channels and chambers that allow for the separation of sperm based on their motility and morphology. The chip is designed to mimic the natural environment of the female reproductive tract, where sperm undergo a series of selection processes before reaching the egg.
  Interventions: Device: Microfluidic chip
- density-gradient centrifugation method (Active Comparator): Density-gradient centrifugation is a commonly used method for sperm separation and purification. It is a technique that involves layering a semen sample on top of a gradient of different densities of a solution, typically a mixture of colloidal silica and sucrose, and then centrifuging the sample. The centrifugal force causes the sperm to migrate through the gradient, where they become separated based on their density.
  Interventions: Device: Density-gradient centrifugation

INTERVENTIONS:
Device: Microfluidic chip — The Sperm Separation Device - ZyMōt Multi 850µL (ZyMōt Fertility, Inc) will be used. The microfluidics chamber will be used according to the manufacturer's instructions. 850 μL of the semen sample will be inserted into the inlet port of the device and 750 μL of fertilization media will be inserted into the outlet port. The device with the semen sample inside will be incubated in 6% CO2 at 37°C. After 30 min, 500 μL of the sample at the outlet port will be removed from the outlet port and pipetted into a labelled test tube.
  Arms: microfluidic chip method
Device: Density-gradient centrifugation — After liquefaction, sperm preparation will be completed by a discontinuous density gradient centrifugation method, using Pureception (CooperSurgical, Denmark) sperm density gradient media. The resulting sperm pellet after centrifugation will be washed once with the sperm washing medium (G-IVF Plus, Vitrolife, Sweden) The washed spermatozoa will be resuspended with the same medium, adjusting the final volume to 0.5 mL.
  Arms: density-gradient centrifugation method

SUMMARY:
Infertile patients attending IVF treatment at the Centre of Assisted Reproduction and Embryology, Queen Mary Hospital and Kwong Wah Hospital will be recruited during ovarian stimulation for IVF. Subsequently, they will be randomly assigned on the day of oocyte retrieval by a laboratory staff into one of the following two groups: (1) the microfluidic chip group and (2) the density gradient group for sperm preparation and subsequent use in fertilization. Other IVF procedures will be the same as our usual practice. Both patients and clinicians were blinded from the group allocation i.e. a double blind study. The primary outcome is the cumulative live birth rate defined as the number of pregnancies leading to live birth within 6 months of randomisation.

DETAILED DESCRIPTION:
The trial will compare the use of a microfluidic chip with the use of density gradient centrifugation for sperm preparation.

The hypothesis of the study is that the use of the microfluidic chip will improve the cumulative live birth rate of IVF compared to the density gradient method.

The trial will be conducted at the Centre of Assisted Reproduction and Embryology at Queen Mary Hospital and Kwong Wah Hospital. Infertile patients undergoing IVF treatment will be recruited during ovarian stimulation. They will be randomly assigned to one of two groups: the microfluidic chip group or the density gradient group. Both the patients and the clinicians will be blinded to the group allocation.

The inclusion criteria for the study are infertile women aged under 43 years undergoing ovarian stimulation for IVF. The exclusion criteria include women undergoing certain genetic testing, male factor infertility requiring surgical sperm retrieval, the use of donor oocytes and spermatozoa, certain uterine conditions, previous participation in the study, and participation in other randomized trials.

The eligible women will undergo standard IVF procedures, including ovarian stimulation, monitoring of follicle growth, trigger for oocyte retrieval, and oocyte retrieval itself. On the day of oocyte retrieval, the women will be randomly assigned to either the microfluidic chip group or the density gradient group for sperm preparation.

Semen samples will be collected on the day of oocyte retrieval and evaluated according to standard guidelines. Sperm DNA damage will also be assessed using an alkaline single-cell gel electrophoresis assay. Depending on the randomization, the sperm samples will be prepared either using the microfluidic chip or the density gradient centrifugation method.

After sperm preparation, oocytes will be fertilized using either conventional insemination or intracytoplasmic sperm injection. Fertilization will be confirmed by the presence of two pronuclei. Fresh embryo transfer will be performed 2-5 days after egg retrieval, and luteal phase support will be given. Excessive good quality embryos or blastocysts will be cryopreserved for future use.

For frozen embryo transfer, embryos or blastocysts will be replaced in subsequent natural or hormonal replacement cycles. Pregnancy will be confirmed by a urine pregnancy test, and transvaginal ultrasound will be performed to confirm viability and the number of fetuses.

Follow-up will be conducted to retrieve pregnancy and delivery data. The cumulative live birth rate will be calculated, and pregnancy outcomes, including birth weights and obstetric complications, will be recorded and compared between the two groups.

The study will continue until all cryopreserved embryos or blastocysts are used or until the participants become pregnant within 6 months after randomization. The pregnancy complications and congenital abnormalities will be monitored through hospital records or patient contact.

Ultimately, the study aims to determine whether the use of the microfluidic chip improves the cumulative live birth rate of IVF compared to the density gradient method.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women aged <43 years at the time of ovarian stimulation for IVF

Exclusion Criteria:

* Women undergoing preimplantation genetic testing monogenic diseases, structural rearrangement of chromosomes or aneuploidy;
* Male factor requiring surgical sperm retrieval such as microscopic epididymal sperm aspiration and testicular sperm extraction;
* Use of donor oocytes and spermatozoa;
* Submucosal fibroid or hydrosalpinx shown on pelvic scanning and not surgically treated;
* Women who had been recruited into this study before and
* Women joining other randomized trials

Max Age: 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1136 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
cumulative live birth rate | within 6 months of randomisation.
  cumulative live birth rate defined as the number of pregnancies leading to live birth within 6 months of randomisation.

SECONDARY OUTCOMES:
Live birth beyond 22 weeks of gestation per the first embryo transfer or FET | 3 years
  Live birth beyond 22 weeks of gestation per the first embryo transfer or FET
Positive urine pregnancy test per the first embryo transfer or FET | 3 years
  Positive urine pregnancy test per the first embryo transfer or FET
Clinical pregnancy per the first embryo transfer or FET defined as presence of intrauterine gestational sac on scanning at gestational week 6. | 3 years
  Clinical pregnancy per the first embryo transfer or FET defined as presence of intrauterine gestational sac on scanning at gestational week 6.
Ongoing pregnancy rate as presence of a fetal pole with pulsation at 8-10 weeks of gestation | 3 years
  Ongoing pregnancy rate as presence of a fetal pole with pulsation at 8-10 weeks of gestation
Miscarriage defined as a clinically recognized pregnancy loss before the 22 weeks of pregnancy and whose denominator is the clinical pregnancy. | 3 years
  Miscarriage defined as a clinically recognized pregnancy loss before the 22 weeks of pregnancy and whose denominator is the clinical pregnancy.
Multiple pregnancy: presence of more than one intrauterine sac at 6 weeks of gestation | 3 years
  Multiple pregnancy: presence of more than one intrauterine sac at 6 weeks of gestation
Ectopic pregnancy rate | 3 years
  Ectopic pregnancy rate

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynaecology, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after publication of the primary paper
Access Criteria: reasonable request